CLINICAL TRIAL: NCT07260604
Title: Randomized Trial on Pelvic Floor Training With and Without HIFEM for Stress Urinary Incontinence
Brief Title: HIFEM for Incontinence After Menopause High-Intensity Focused Electromagnetic (HIFEM)
Acronym: HIM2025
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FoU in Sweden 284879
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Urinary Incontinence (UI)
Keywords: urinary incontinence; pelvic floor training; HIFEM-treatment
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Before the RCT, a case study will be performed. In addition, a qualitative study part is included in the RCT
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor) - physiotherapist performing muscle strength assessment blinded to allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Standard Pelvic Floor Training (Active Comparator): * Active pelvic floor muscle training led by a physiotherapist, following standard practice.
  * Includes individualized advice and daily Kegel exercises to increase endurance and strength.
  Interventions: Other: Pelvic Floor exercises
- Arm B - Pelvic Floor Training + HIFEM (Experimental): * Same physiotherapist-led training as Arm A.
  * In addition: HIFEM treatment with Emsella chair.
  * 10 sessions, 30 min each, over 5 weeks (2 sessions per week).
  * Standardized stimulation delivered while seated, fully clothed, in a nurse-led clinic in Gothenburg.
  Interventions: Device: Pelvic floor training as described in point a above, with the addition of HIFEM.

INTERVENTIONS:
Device: Pelvic floor training as described in point a above, with the addition of HIFEM. — Pelvic floor training with the addition of HIFEM. The treatment will be administered over 8-10 sessions of 30 minutes each, over a period of 4-6 weeks, with two sessions per week. During treatment, the women will sit fully clothed in a treatment chair and receive standardized stimulation of the pelvic floor muscles.
  Arms: Arm B - Pelvic Floor Training + HIFEM
Other: Pelvic Floor exercises — Pelvic floor training according to national guidelines
  Arms: Arm A - Standard Pelvic Floor Training

SUMMARY:
It is not difficult to imagine that leaking urine affects life in many contexts. Unfortunately, it is everyday life for far too many people in our society. According to the National Board of Health and Welfare, incontinence primarily affects older people, and both women and men are vulnerable. In Sweden, just over 530,000 people over the age of 65 have problems and almost 80 percent of all people in special housing have such urine leakage that they need to use incontinence aids. First-line treatment for women with incontinence is local estrogen and pelvic floor training. Surgery may also be considered if this treatment does not provide sufficient effect.

A new type of treatment for stress, urge and mixed incontinence is now on the market, High-Intensity Focused Electromagnetic (HIFEM®) treatment. This involves electromagnetic stimulation that causes contractions in the pelvic floor muscles. The treatment is not painful or invasive and the patient sits clothed in the treatment chair. In Sweden, HIFEM® is mainly available outside of traditional healthcare and is very expensive. It is also often given by unauthorized actors.

We are now planning a study whose purpose is to evaluate the effect of HIFEM® on women over 65 years of age with stress incontinence. A group of 100 women will be randomized to:

1. Standard treatment, i.e. physiotherapy-led pelvic floor training
2. As above with the addition of 10 treatments of 30 minutes with HIFEM®.

The evaluation will be carried out regarding leakage, need for incontinence aids and pelvic floor strength immediately and six months after the intervention. The women will also rate their incontinence symptoms, physical activity level, physical function and quality of life. A group will also be interviewed about their experiences of living with incontinence and the treatment. Before the study start, a case study will be performed in which 10 women will be included. They will receive 10 treatments and measure, with the same outcomes, the effects.

Alternative treatment methods are important to meet the care needs we have today but also in the future. If treatment with HIFEM® can be effective for women over 65, it could, in addition to reducing incontinence problems and the consequences of these problems, also lead to reduced costs for society regarding care and incontinence products, as well as reduced environmental impact.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 65-85 ears
* Having daily stress incontinence requiring use of incontinence aids.
* Living in ordinary housing without home (health-) care
* Being physically active and can move independently both indoors and outdoors.
* Being able to give independent informed consent in speech and writing
* To understand and follow instructions in one of following languages Swedish, Arabic, French, and/or English

Exclusion Criteria:

* -Ongoing coached pelvic floor training
* Heart disease where treatment is contraindicated
* Lung disease with chronic cough
* Pacemaker, defibrillator, neurostimulator, medication pump, and implanted devices in the head or spinal cord
* Electronic or metal implants in the abdomen, hips, or knees
* Epilepsy
* Ongoing cancer
* Stoma or abdominal hernia
* Ongoing treatment with anticoagulants such as warfarin, medicines affecting the bladder such as muscarin receptor antagonist, diuretics and local oestrogen which affect the bladder and urine production.
* infection, fever, bleeding, or pain in the lower abdomen
* Skin diseases or any skin sensitivity
* BMI exceeding 30 kg/m2

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Women, aged 65-85 years.
Enrollment: 100 (Estimated)
Dates: Start 2026-10-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Leakage volume | From enrollment to the end of treatment at 5 weeks. Follow up at 6 months and at 1 year.
  Weight of leakage
Urinary incontinence severity | Baseline, post-treatment, 6 months, 12 months
  International Consultation on Incontinence Questionnaire-short form ICIQ-SF.

SECONDARY OUTCOMES:
Number of leakage/day | From enrollment to the end of treatment at 5 weeks. Follow up at 6 months and at 1 year.
  Number/ day
Need of continence aids | From enrollment to the end of treatment at 5 weeks. Follow up at 6 months and at 1 year.
  Number of aids used per day
Pelvic floor muscle strength | Before and after the intervention
  Modified Oxford Scale, pre- and post-treatment, blinded assessor
Impact of urinary incontinence on sexual health | At baseline, post-treatment, 6 months, and 12 months.
  The questionnaire "Impact of urinary incontinence on sexual health (ICIQ-FLUTSsex)."
Health-related quality of life | At baseline, post-treatment, 6 months, and 12 months.
  Questionnaire: Pelvic Floor Impact Questionnaire - Short Form 7 (PFIQ-7) som
Rated physical function | At baseline, post-treatment, 6 months, and 12 months
  Patient-Specific Functional Scale (PSFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg university, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No